CLINICAL TRIAL: NCT00002121
Title: Diethylhomospermine (DEHSPM) for Refractory AIDS-Related Diarrhea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Medical Center-Gainesville (U.S. Federal Agency)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 223A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Diarrhea; HIV Infections
Keywords: Antidiarrheals; Diarrhea; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; N(1),N(14)-bis(ethyl)homospermine
MeSH Terms: conditions — Diarrhea; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — N(1),N(14)-bis(ethyl)homospermine

INTERVENTIONS:
Drug: Diethylhomospermine

SUMMARY:
To perform preliminary clinical testing of diethylhomospermine (DEHSPM), a polyamine analogue, for refractory AIDS-related diarrhea.

Possibly, DEHSPM will reduce stool volume and frequency in patients with refractory AIDS-related diarrhea.

DETAILED DESCRIPTION:
Possibly, DEHSPM will reduce stool volume and frequency in patients with refractory AIDS-related diarrhea.

Patients are initially hydrated for 24 hours, followed by a 3-day baseline period. They then receive intravenous infusions of DEHSPM three times per day for 3 days, followed by observation for 3 days.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* ARC or AIDS by CDC criteria.
* Uncontrolled diarrhea unresponsive to high-dose, nonspecific antidiarrheal therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known idiopathic ulcerative colitis or Crohn colitis.
* Acute stool-culture-positive bacterial colitis.
* Acute amoebic colitis.
* Pseudomembranous colitis with Clostridium difficile toxin positivity.
* Short-gut syndrome.
* Chronic pancreatitis.
* Ischemic bowel disease.
* Enteroenteric fistulae.
* Other gastrointestinal tract disorders known to cause diarrhea.
* Underlying evidence of immunosuppression other than that related to HIV infection.
* Unable or unwilling to have subcutaneous injections.
* Clinically significant CNS, hepatic, or renal disease.

Concurrent Medication:

Excluded:

* Other experimental antidiarrheal drugs.
* Antibiotic therapy.

Prior Medication:

Excluded:

* Other experimental drugs within 1 month prior to study entry.

Required:

* At least 2 weeks of prior high-dose, nonspecific antidiarrheal therapy (i.e., loperamide, diphenoxylate hydrochloride-atropine sulfate, or opiates) at maximally tolerable doses.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Gainesville Veterans Administration Med Ctr, Gainesville, Florida, United States